CLINICAL TRIAL: NCT02598791
Title: GIP/GLP-1 Co-Activity in Subjects With Obesity: Lowering of Food Intake
Acronym: GASOLIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Natasha Chidekel Bergmann, MD Ph.D student, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-15008790 (GASOLIN)
Record Dates: First submitted 2015-10-31; First posted 2015-11-06 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Obesity; Adiposity; Type 2 Diabetes
Keywords: incretin hormones; GIP; GLP-1
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- IIGI+GIP (Active Comparator): 4 hour i.v. infusion of glucose-dependent insulinotropic polypeptide (4 pmol/kg/min) during isoglycemic conditions
  Interventions: Other: IIGI+GIP; Other: IIGI+GLP-1; Other: IIGI+NaCl (placebo); Other: OGTT; Other: IIGI+GIP+GLP-1
- IIGI+GLP-1 (Active Comparator): 4 hour i.v. infusion of glucagon-like peptide-1 (1 pmol/kg/min) during isoglycemic conditions
  Interventions: Other: IIGI+GIP; Other: IIGI+GLP-1; Other: IIGI+NaCl (placebo); Other: OGTT; Other: IIGI+GIP+GLP-1
- IIGI+NaCl (placebo) (Placebo Comparator): 4 hour i.v. NaCl (placebo) during isoglycemic conditions
  Interventions: Other: IIGI+GIP; Other: IIGI+GLP-1; Other: IIGI+NaCl (placebo); Other: OGTT; Other: IIGI+GIP+GLP-1
- IIGI+GIP+GLP-1 (Active Comparator): 4 hour co-infusion of glucose-dependent insulinotropic polypeptide and glucagon-like peptide-1
  Interventions: Other: IIGI+GIP; Other: IIGI+GLP-1; Other: IIGI+NaCl (placebo); Other: OGTT; Other: IIGI+GIP+GLP-1
- 50 g OGTT (Other): 50 g oral glucose tolerance test (OGTT)
  Interventions: Other: IIGI+GIP; Other: IIGI+GLP-1; Other: IIGI+NaCl (placebo); Other: OGTT; Other: IIGI+GIP+GLP-1

INTERVENTIONS:
Other: IIGI+GIP — Glucose-dependent insulinotropic polypeptide (4 pmol/kg/min) during isoglycemia
Other: IIGI+GLP-1 — glucagon-like peptide-1 (1 pmol/kg/min) during isoglycemia
Other: IIGI+NaCl (placebo) — i.v. NaCl during isoglycemia
Other: OGTT — 50 g oral glucose tolerance test
Other: IIGI+GIP+GLP-1 — i.v infusion of GIP and GLP-1 (4 + 1 pmol/kg/min) during isoglycemia

SUMMARY:
We aim to delineate the effects of separate and combined infusion of GIP and GLP-1 on food intake, appetite, bone health and fat metabolism in overweight/obese subjects.

DETAILED DESCRIPTION:
The gut-derived incretin glucagon-like peptide-1 (GLP-1) is a potent regulator of gastric emptying, appetite and food intake in humans whereas its sister incretin hormone, glucose-dependent insulinotropic polypeptide (GIP), does not seem to have independent effects on these variables in humans. Interestingly, recent data from rodents have shown that concomitant activation of the GIP and the GLP-1 receptor may potentiate the satiety-promoting and body weight-reducing effects of GLP-1. Also, evidence suggests that GIP may be an important mediator of bone remodelling and lipid deposition. The effect of simultaneous activation of the GIP and GLP-1 receptors on appetite, food intake, fat metabolism and bone health has not been thoroughly examined in humans. The aim of this study is to delineate the effects of GIP/GLP-1 receptor co-activation on food intake, mechanisms regulating food intake, fat and bone metabolism in obese subjects.

Material and methods:

The investigators plan to include 18 obese/overweight men without diabetes. The primary endpoint of the study is food intake during continuous intravenous infusions of saline (placebo), GIP, GLP-1 and GIP+GLP-1, respectively. Secondary endpoints includes resting energy expenditure (measured by indirect calorimetry), appetite, satiety and hunger assessments (measured by visual analogue scales), plasma insulin, C-peptide and glucagon secretion, plasma triglycerides, cholesterols, and free fatty acid responses and changes in plasma bone turnover markers.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men
* Age between 25 and 70 years
* Body mass index (BMI) between 25 and 40 kg/m2

Exclusion Criteria:

* Diabetes or prediabetes (defined as glycated haemoglobin (HbA1c) ≥ 43 mmol/mol)
* Anaemia (defined as haemoglobin < 8.3 mmol/l)
* Any gastrointestinal disease that may interfere with the endpoint variables
* Anorexia, bulimia or binge eating disorder
* Allergy or intolerance to ingredients included in the standardised meals
* Tobacco smoking
* Any regular drug treatment that cannot be discontinued for minimum 18 hours
* Any physical or psychological condition that the investigator feels would interfere with trial participation

Ages: 25 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
food intake | 250-280 min
  How much does the participant eat of from the ad libitum meal, measured in gram

SECONDARY OUTCOMES:
hunger | measured at time 0, 30, 60, 90, 120, 180, 210, 240 min
  feeling of hunger measured on a visual analogue scale
satiety | measured at time 0, 30, 60, 90, 120, 180, 210, 240 min
  feeling of satiety measured on a visual analogue scale
Fullness | measured at time 0, 30, 60, 90, 120, 180, 210, 240 min
  feeling of fullness measured on a visual analogue scale
Prospective food consumption | measured at time 0, 30, 60, 90, 120, 180, 210, 240 min
  Prospective food consumption measured on a visual analogue scale
resting energy expenditure (REE) | -15 to 0 min. and 210 to 225 min.
  changes in REE measured by a ventilated hood 15 minutes at baseline and 15 minutes at time point 210 min.
Insulin | -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min
  changes in insulin measured in serum
C-peptide level | -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min
  changes in C-peptide level measured in serum
glucagon levels | -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min
  changes in glucagon levels measured in plasma
Cholesterol and FFA | -30, 0, 30, 60, 90, 120, 180, 240 min
  changes in cholesterol (TAG, Total cholesterol and free fatty acid measured in plasma)
C-terminal cross-linked telopeptide of bone collagen (CTX) | -30, 0, 30, 60, 90, 120, 180, 240 min
  changes in level of CTX measured in plasma
procollagen type 1 N-terminal propeptide (P1NP) | -30, 0, 30, 60, 90, 120, 180, 240 min
  changes in level of P1NP measured in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Natasha C Bergmann, MD, Principal Investigator — Center for Diabetesresearch, Gentofte Hospital, University of Copenhagen, Denmark
Locations (1):
- Center for Diabetesresearch, Gentofte hospital, Hellerup, Denmark

REFERENCES:
- [Background] Finan B, Ma T, Ottaway N, Muller TD, Habegger KM, Heppner KM, Kirchner H, Holland J, Hembree J, Raver C, Lockie SH, Smiley DL, Gelfanov V, Yang B, Hofmann S, Bruemmer D, Drucker DJ, Pfluger PT, Perez-Tilve D, Gidda J, Vignati L, Zhang L, Hauptman JB, Lau M, Brecheisen M, Uhles S, Riboulet W, Hainaut E, Sebokova E, Conde-Knape K, Konkar A, DiMarchi RD, Tschop MH. Unimolecular dual incretins maximize metabolic benefits in rodents, monkeys, and humans. Sci Transl Med. 2013 Oct 30;5(209):209ra151. doi: 10.1126/scitranslmed.3007218. PMID 24174327
- [Background] Campbell JE, Drucker DJ. Pharmacology, physiology, and mechanisms of incretin hormone action. Cell Metab. 2013 Jun 4;17(6):819-837. doi: 10.1016/j.cmet.2013.04.008. Epub 2013 May 16. PMID 23684623
- [Background] Flint A, Raben A, Astrup A, Holst JJ. Glucagon-like peptide 1 promotes satiety and suppresses energy intake in humans. J Clin Invest. 1998 Feb 1;101(3):515-20. doi: 10.1172/JCI990. PMID 9449682
- [Background] Nissen A, Christensen M, Knop FK, Vilsboll T, Holst JJ, Hartmann B. Glucose-dependent insulinotropic polypeptide inhibits bone resorption in humans. J Clin Endocrinol Metab. 2014 Nov;99(11):E2325-9. doi: 10.1210/jc.2014-2547. Epub 2014 Aug 21. PMID 25144635
- [Derived] Bergmann NC, Lund A, Gasbjerg LS, Jorgensen NR, Jessen L, Hartmann B, Holst JJ, Christensen MB, Vilsboll T, Knop FK. Separate and Combined Effects of GIP and GLP-1 Infusions on Bone Metabolism in Overweight Men Without Diabetes. J Clin Endocrinol Metab. 2019 Jul 1;104(7):2953-2960. doi: 10.1210/jc.2019-00008. PMID 30848791
- [Derived] Bergmann NC, Lund A, Gasbjerg LS, Meessen ECE, Andersen MM, Bergmann S, Hartmann B, Holst JJ, Jessen L, Christensen MB, Vilsboll T, Knop FK. Effects of combined GIP and GLP-1 infusion on energy intake, appetite and energy expenditure in overweight/obese individuals: a randomised, crossover study. Diabetologia. 2019 Apr;62(4):665-675. doi: 10.1007/s00125-018-4810-0. Epub 2019 Jan 25. PMID 30683945